CLINICAL TRIAL: NCT06782711
Title: Efficacy and Safety of Customized Skull Implants Made of Polyetheretheretherketone Using Three-dimensional Printing in Patients Undergoing Cranioplasty
Brief Title: Efficacy and Safety of 3D-Printed PEEK Skull Implants in Cranioplasty
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: CIMET SCIENTIFIC CORPORATION (Other)
Collaborators: Consejo Nacional de Humanidades, Ciencias y Tecnologias (CONAHCYT) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIMET-2024-01
Record Dates: First submitted 2025-01-08; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Cranial Defects
Keywords: Cranioplasty; Custom implants; Polyetheretheretherketone (PEEK); Three-dimensional (3D) printing; Neurosurgery; Cranial prostheses; Medical devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cranioplasty using customized skull implants made of polyetheretheretherketone using 3D printing (Experimental): All participants will undergo cranioplasty using customized skull implants made of polyetheretheretherketone using 3D printing
  Interventions: Procedure: cranioplasty; Device: customized skull implants made of polyetheretheretherketone (PEEK) using 3D printing

INTERVENTIONS:
Procedure: cranioplasty — In this pivotal study of a medical device, patients with bone loss undergo a computed tomography scan, which is used to create a three-dimensional model of the lesion. After validation, the model is printed using PEEK material, and subsequently, the skull is repaired through cranial reconstruction (cranioplasty).
Device: customized skull implants made of polyetheretheretherketone (PEEK) using 3D printing — customized skull implants made of polyetheretheretherketone by three-dimensional printing in patients undergoing cranioplasty

SUMMARY:
The goal of this clinical trial is to determine the efficacy and safety of customized skull implants made of polyetheretheretherketone by three-dimensional printing in patients undergoing cranioplasty. The main question it aims to answer is:

• Are customized skull implants made of polyetheretheretherketone using 3D printing effective and safe in patients undergoing cranioplasty?

Participants will:

* The patient will be submitted to cranioplasty.
* The patient will answer the neurological scales at each visit.
* Keep a diary of their symptoms and concomitant medications
* The study will be divided into 5 visits to the center, the surgical intervention and 3 telephone calls where patients will be followed up.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy and safety of personalized skull implants made of polyetheretheretherketone (PEEK) using three-dimensional printing in patients undergoing cranioplasty. This is a phase II clinical trial, with a single group of 30 patients who have suffered cranial bone loss. Specific objectives include analyzing the incidence of complications (infections, fractures, implant exposure), assessing functional recovery using recognized scales such as the Glasgow and Barthel scales, and measuring patient and surgeon aesthetic satisfaction over 12 months.

The design includes multiple follow-up visits, from surgery to one year after, where neurological, functional and cosmetic assessments will be performed.

The selection and exclusion criteria ensure the suitability of the participants, while the variables monitored allow a comprehensive analysis of the results, from cognitive functionality to surgical complications. This study seeks to provide scientific evidence to support the implementation of this technology in patients with cranial defects, improving both quality of life and post-surgical aesthetic and functional outcomes.

-Main inclusion criteria: Being older than 18 years, of both sexes. Loss of cranial bone segment greater than 1 cm². Glasgow Coma Scale (GCS) score equal or greater than 9. Satisfactory pre-surgical evaluation. Signed informed consent.

-Main exclusion criteria: Local infection at the craniotomy site or active systemic infection. Presence of previous surgical instruments at the cranioplasty site. Need to use two or more implants for reconstruction. History of coagulopathies, uncontrolled diabetes mellitus or body mass index (BMI) greater than 35.

Pregnant or lactating women.

-Main variables: Efficacy and safety: frequency of complications such as infections, fractures and implant exposure.

Cognitive functionality: Assessed by the Mini-Mental State Examination (MMSE). Functional independence: Measured with the Barthel index. Degree of disability: Assessed with the Modified Rankin Scale (mRS). Cosmetic satisfaction: Patient and surgeon satisfaction. Adverse events: Incidence during the 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old.
* Both sexes.
* Who agree to participate and sign the informed consent form.
* With loss of a bone segment.
* Area of bone segment loss greater than 1 cm.
* Glasgow Coma Scale score equal to or greater than 9.
* Satisfactory preoperative evaluation

Exclusion Criteria:

* Presence of local infection at the craniotomy site or any type of systemic infection at the time of medical evaluation and systemic infection at the time of medical evaluation and during surgery.
* Presence of previous surgical instruments in the cranioplasty site.
* Need to use two or more implants for the reconstruction.
* The resulting angle between the tangential lines to the curvature of the implant and the tangent determined to the center of the implant, determined to the center of the implant, is greater than 50º.
* Patients whose cranial morphology presents difficulties for the prosthesis design.
* Presence of postoperative ossifications in the defect area.
* History of hypersensitivity to biomaterials.
* Surgery at the same site within the 6 months prior to the study surgery.
* Patients with any diagnosis that affects blood supply and bone quality.
* Patients who have received chemotherapy or radiotherapy in the surgical region that ended within 6 months prior to the planned surgery or are scheduled for the next 12 weeks.
* Diagnosis of malignant cranial tumor.
* History of any status epilepticus.
* Known history of hemophilia or other clinically significant coagulopathy.
* Patients with uncontrolled diabetes according to, ADA criteria:

  o fasting glucose ≥ 200 mg/dL, HbA1C ≥ 8.5% in the last 3 months.
* Patients with a body mass index (BMI) ≥ 35 kg/m
* History of steroid drugs at least 3 months before surgery.
* Women breastfeeding or pregnant.
* Inability to read and understand the participant's information.
* Prior participation in any related investigational drug or device study within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Frequency and causes of cranioplasty revisions | From enrollment to the end of treatment at 12 months
  Cranioplasty revision is performed when it is necessary to correct or adjust a previously placed implant, either due to complications adjust a previously placed implant, either due to complications, lack of integration of the implant or changes in the desired form and function.

SECONDARY OUTCOMES:
Infection at the implant site | From enrollment to 3 months after surgery
  Evaluate the frequency of infection at the implant site after cranioplasty.
Frequency of surgery-associated infections | From enrollment to 3 months after surgery
  These are infections that develop as a direct result of a surgical procedure. These infections can affect various parts of the body and are not necessarily limited to the implant site.
Frequency of implant exposure | From enrollment to the end of treatment at 12 months
  It refers to the fact that the implants placed in the cranial region, in reconstructive or reparative surgeries of the skull, are visible or accessible in some way.
Frequency and type of implant fractures | From enrollment to the end of treatment at 12 months
  Refers to the rupture or cracking of devices implanted in the cranial region, used in reconstructive or reparative surgeries of the skull.
Level of consciousness | From enrollment to 3 months after surgery
  Establish the level of consciousness with the Glasgow Coma Scale (GCS).
Cognitive function | From enrollment to the end of treatment at 12 months
  Measure cognitive function with the Mini-Mental State Examination (MMSE).
Functional independence | From enrollment to the end of treatment at 12 months
  Evaluate functional independence with the Barthel Index.
Level of disability | From enrollment to the end of treatment at 12 months
  Evaluate the degree of disability with the modified Rankin Scale (mRS).
Cosmetic satisfaction | From enrollment to the end of treatment at 12 months
  Subjective scale to assess patient and surgeon satisfaction in terms of aesthetic and functional results after cranioplasty surgery.
Frequency of adverse incidents | From enrollment to the end of treatment at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Geannyne Villegas Rivera, MD, PhD, MBA, Study Director — Centro de Investigación Clínica y Medicina Traslacional (CIMET)
Locations (1):
- Centro de Investigación Clínica y Medicina Traslacional (CIMET), Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share IPD is currently 'Undecided' because further discussions and evaluations are needed regarding the feasibility, ethical considerations, and alignment with institutional policies. Once these factors are thoroughly assessed, a final determination will be made.

REFERENCES:
- [Background] Yang J, Sun T, Yuan Y, Li X, Yu H, Guan J. Evaluation of titanium mesh cranioplasty and polyetheretherketone cranioplasty: protocol for a multicentre, assessor-blinded, randomised controlled trial. BMJ Open. 2019 Dec 3;9(12):e033997. doi: 10.1136/bmjopen-2019-033997. PMID 31796495
- [Background] Sharma N, Aghlmandi S, Dalcanale F, Seiler D, Zeilhofer HF, Honigmann P, Thieringer FM. Quantitative Assessment of Point-of-Care 3D-Printed Patient-Specific Polyetheretherketone (PEEK) Cranial Implants. Int J Mol Sci. 2021 Aug 7;22(16):8521. doi: 10.3390/ijms22168521. PMID 34445228
- [Background] Mozaffari K, Rana S, Chow A, Mahgerefteh N, Duong C, Sheppard JP, Phillips HW, Jarrahy R, Yang I. Customized polyetheretherketone (PEEK) implants are associated with similar hospital length of stay compared to autologous bone used in cranioplasty procedures. J Neurol Sci. 2022 Mar 15;434:120169. doi: 10.1016/j.jns.2022.120169. Epub 2022 Jan 24. PMID 35134672
- [Background] Henry J, Amoo M, Taylor J, O'Brien DP. Complications of Cranioplasty in Relation to Material: Systematic Review, Network Meta-Analysis and Meta-Regression. Neurosurgery. 2021 Aug 16;89(3):383-394. doi: 10.1093/neuros/nyab180. PMID 34100535
- [Background] Csamer L, Csernatony Z, Novak L, Kovari VZ, Kovacs AE, Soosne Horvath H, Mano S. Custom-made 3D printing-based cranioplasty using a silicone mould and PMMA. Sci Rep. 2023 Jul 25;13(1):11985. doi: 10.1038/s41598-023-38772-9. PMID 37491550
- [Background] Basgul C, Yu T, MacDonald DW, Siskey R, Marcolongo M, Kurtz SM. Structure-Property Relationships for 3D printed PEEK Intervertebral Lumbar Cages Produced using Fused Filament Fabrication. J Mater Res. 2018 Jul 27;33(14):2040-2051. doi: 10.1557/jmr.2018.178. Epub 2018 Jun 18. PMID 30555210
- [Background] Alkhaibary A, Alharbi A, Alnefaie N, Oqalaa Almubarak A, Aloraidi A, Khairy S. Cranioplasty: A Comprehensive Review of the History, Materials, Surgical Aspects, and Complications. World Neurosurg. 2020 Jul;139:445-452. doi: 10.1016/j.wneu.2020.04.211. Epub 2020 May 6. PMID 32387405